CLINICAL TRIAL: NCT06406270
Title: Alternative Protein Short Chronic Study
Acronym: APSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: University of Aberdeen
Record Dates: First submitted 2023-11-20; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fava-based diet (Experimental): At the end of the morning of each intervention visit, participants were provided with meals, which they consumed for seven consecutive days (in a 4-day rotation menu). Participants were instructed to consume only the meals that were provided to them during the study days. The breakfast, lunch and dinner meals of the diets were designed to contain 30% fat, 15% protein, 55% carbohydrate, and seven different menus (1500, 1750, 2000, 2250, 2500, 2750 and 3000 Kcal) to deliver the closest energy requirements of the volunteers. For the intervention diets, all the meat was replaced with buckwheat and fava bean food products, serving the same amount of buckwheat and fava bean food products for all the volunteers regardless of their energy requirements.
  Interventions: Other: Fava
- Buckwheat-based diet (Experimental): At the end of the morning of each intervention visit, participants were provided with meals, which they consumed for seven consecutive days (in a 4-day rotation menu). Participants were instructed to consume only the meals that were provided to them during the study days. The breakfast, lunch and dinner meals of the diets were designed to contain 30% fat, 15% protein, 55% carbohydrate, and seven different menus (1500, 1750, 2000, 2250, 2500, 2750 and 3000 Kcal) to deliver the closest energy requirements of the volunteers. For the intervention diets, all the meat was replaced with buckwheat and fava bean food products, serving the same amount of buckwheat and fava bean food products for all the volunteers regardless of their energy requirements.
  Interventions: Other: Buckwheat

INTERVENTIONS:
Other: Fava — Participants were instructed to consume only the meals that were provided to them during the study days. The breakfast, lunch and dinner meals of the diets were designed to contain 30% fat, 15% protein, and 55% carbohydrate, and seven different menus (1500, 1750, 2000, 2250, 2500, 2750 and 3000 Kcal) to deliver the closest energy requirements of the volunteers. For the intervention diets, all the meat was replaced with fava bean food products, serving the same amount of buckwheat and fava bean food products for all the volunteers independently of their energy requirements. During the intervention diets, all the drinks, such as coffee, juice and tea, were restricted and provided by the Human Nutrition Unit at the Rowett Institute; the volunteers were allowed to drink only water ad libitum. Alcoholic drinks were not allowed to be consumed during the intervention diet weeks.
  Arms: Fava-based diet
Other: Buckwheat — Participants were instructed to consume only the meals that were provided to them during the study days. The breakfast, lunch and dinner meals of the diets were designed to contain 30% fat, 15% protein, and 55% carbohydrate, and seven different menus (1500, 1750, 2000, 2250, 2500, 2750 and 3000 Kcal) to deliver the closest energy requirements of the volunteers. For the intervention diets, all the meat was replaced with buckwheat food products, serving the same amount of buckwheat and fava bean food products for all the volunteers independently of their energy requirements. During the intervention diets, all the drinks, such as coffee, juice and tea, were restricted and provided by the Human Nutrition Unit at the Rowett Institute; the volunteers were allowed to drink only water ad libitum. Alcoholic drinks were not allowed to be consumed during the intervention diet weeks.
  Arms: Buckwheat-based diet

SUMMARY:
The world's population needs adequate food supply to sustain food security. The availability of sufficient dietary protein is undeniably a source of concern for human health. This study aimed to assess the satiety and potential health benefits of two types of vegetarian diets when the meat was replaced with buckwheat and respectively fava bean for one-week in the diet of healthy volunteers.

DETAILED DESCRIPTION:
The World Health Organisation (WHO) recommends increasing the intake of fruits and vegetables, legumes, whole grains and nuts to prevent obesity. In Western countries, there is a greater understanding of the health benefits of pulse grains. Consumption of whole grain cereals and grain pulses has been shown to protect against a variety of inflammation-related chronic diseases. Grain cereals, pulses and pseudo cereals are also good dietary protein sources. This study aimed to assess the suitability of buckwheat and fava bean to replace meat for one week in terms of delivering adequate nutrient intake, satisfying hunger and delivering potential health benefits. The composition of human microbial metabolites and the bacterial composition after consumption of the intervention diets by healthy volunteers for one week were also assessed. This study offers data to support the potential of plants as alternative sources of dietary nutrients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females,
* Non-vegetarian,
* non-smokers,
* age 18-65
* with BMI 18-35 kg/m.

Exclusion criteria:

* vegetarian,
* smoker,
* having known allergies,
* using prescription drugs.
* diabetes,
* gastrointestinal disorders,
* kidney disease,
* hepatic disease,
* favism,
* alcohol or
* substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
The suitability of a vegetarian diet (buckwheat and fava bean based) to deliver sufficient nutrients per day | 7-days
  The suitability of a vegetarian diet (buckwheat and fava bean based) to deliver sufficient nutrients per day such as protein composition, amino acids composition, fibre composition, types of NSP, and daily requirements minerals, microelements, and other bioactive such as polyphenolic phytochemicals. The macronutrient composition, including the dry matter, ash, fat, total carbohydrate, resistant starch, crude protein, and total non-starch polysaccharides of the buckwheat and fava-bean diets are measured in grams per day. The amino acid composition was measured in grams per day and the main micronutrients expressed in mg ± SD per day are measured in fava bean and buckwheat diets using quantitative ICP-MS analysis.
Satiety levels following the consumption of buckwheat and fava bean-based diets. | every hour for 16 hours during the day for 7 days
  Appetite scores were measured hourly during the waking hours (0700-2300) with the use of visual analogue scales (VASs) during both the habitual diet week and the intervention weeks (fava bean-based and buckwheat-based diets). Six questions were asked on motivation to eat, all in the line scale format related to hunger, thirst, preoccupation with thoughts of food, fullness, desire to eat, and prospective consumption. The scales ranged from "not at all hungry" to "extremely hungry," so higher scores indicated more intense subjective sensations. These questionnaires were completed by the subjects each day of the study.
Hourly hunger scores analysed using VAS | every hour for 16 hours during the day for 7 days
  Hunger scores were measured hourly during the waking hours (0700-2300) with the use of visual analogue scales (VASs) during both the habitual diet week and the intervention weeks (fava bean-based and buckwheat-based diets). Six questions were asked on motivation to eat, all in the line scale format related to hunger, thirst, preoccupation with thoughts of food, fullness, desire to eat, and prospective consumption. The scales ranged from "not at all hungry" to "extremely hungry," so higher scores indicated more intense subjective sensations. These questionnaires were completed by the subjects each day of the study.
Concentrations of plasma, urine, and faecal samples of microbial metabolites of carbohydrates, protein, and bioactive phytochemicals. | Baseline and day 7
  Concentrations of plasma, urine, and faecal samples of microbial metabolites of carbohydrates, protein and bioactive phytochemicals from the diets at day 0 and day 7 in fasted plasma, urine and faecal samples. Furthermore looked at fermentation products of carbohydrates in faecal samples. Average concentration was measured by targeted LC-MS/MS and expressed as pg/μl.
Gut microbiota composition: Bacterial DNA extraction and sequencing using 16sRNA to determine the bacterial composition following the two different vegetarian-based diets. | 7-days
  The total number of 16S rRNA gene copies per ml and abundance of several bacterial genera or species of the communities in the anaerobic faecal incubation experiments was determined by quantitative PCR with 2 ng DNA in a total volume of 10 μl and expressed as 16S rRNA gene copies per ml of culture. The abundance of total faecal microbiota and specific genera were reported during habitual (baseline) diet and intervention diets consumption.

SECONDARY OUTCOMES:
Values concentration (μM) of fasted homocysteine | 7-days
  Blood was collected directly into heparinised tubes at day 0 and 7 of each intervention diet. Homocysteine was expressed as μM.
Values concentration (mmol/l) of fasted lipids, urea, and glucose | 7-days
  Blood was collected directly into heparinised tubes at day 0 and 7 of each intervention diet. Fasted lipids, urea and glucose were expressed as mmol/l.
Values concentration (pmol/l) of fasted insulin | 7-days
  Blood was collected directly into heparinised tubes at day 0 and 7 of each intervention diet. Insulin was expressed as pmol/l.

IPD SHARING:
Plan to Share IPD: No